CLINICAL TRIAL: NCT02252757
Title: Validation of Measurements From CoVa Sensor (VALIDATION-CO-1) Study to Assess Measurements of Wireless Cardiac Output Device
Brief Title: Assess Measurements of Wireless Cardiac Output Device
Acronym: Remote-CO-1
Status: Completed | Type: Observational
Sponsor: Aventyn, Inc. (Industry)
Collaborators: Baxter Healthcare Corporation (Industry); BMS Hospital Trust (Other); Intel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: AV.CO.v0-01
Record Dates: First submitted 2014-09-20; First posted 2014-09-30 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Congestive Heart Failure
Keywords: mHealth, hypertension, atherosclerotic disease, diabetes, obesity, metabolic syndrome, cardiotoxins, cardiomyopathy, dsypnea
MeSH Terms: conditions — Heart Failure; Hypertension; Diabetes Mellitus; Obesity; Metabolic Syndrome; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CoVa
  Other Names: Vitalbeat Remote Disease Managment

SUMMARY:
Heart failure is a common cardiovascular problem which is increasing in both prevalence and incidence and associated with substantial morbidity and mortality. The management of heart failure patients is complex and has become a priority world over. Effective methods to keep heart failure patients out of the hospital are essential, both in the interests of the patient's health, as well as to reduce the burden on the health care system

DETAILED DESCRIPTION:
Heart failure patients should be in a position to provide readings of their weight, blood pressure, fluid intake, thoracic fluid, heart rate, heart rate variability, respiration rate, stroke volume, cardiac output, medications and other important parameters and communicate this data to care providers using wireless technology. This data should be made available to medical personnel regularly and on a periodic basis. In this manner the health care providers can detect and respond to warning signs or alerts before the patient's condition worsens to warrant a visit to the doctor or a hospital admission with features of heart failure decompensation. Programs for chronic heart failure that include remote monitoring have been shown to have a positive effect on clinical outcomes in community dwelling patients with chronic heart failure.

In preparation for a study evaluating the effectiveness of mobile monitoring, the value of Stroke Volume and Cardiac Output need to be validated against FDA approved devices that are available in a hospital or clinic setting. This study covers the validation of the measurements taken with the proposed home monitoring device, Perminova's CoVaTM Sensor (Sensor) against clinic devices such as bio-impedance devices, echocardiogram, Doppler and/or MRI

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender above the age of 18 years
* The subject is able and willing to provide written informed consent prior to enrollment in the study
* One or more of the following diagnosis
* New York Heart Association (NYHA) classification class of I-IV or Stages A-D
* Symptoms of dyspnea
* Chronic renal failure on renal replacement therapy

Exclusion Criteria:

* Patients who may not come for follow up or likely to drop out of the study
* Any illness which may preclude regular follow up
* Patient is unable or not willing to wear electrode patches as required
* Patient has skin sensitivity to adhesive or hydrogel materials used in electrode patches
* Patient is considered by the PI to be medically unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is targeted towards at-risk heart failure patients. An "at-risk" patient is defined as a patient who has risk factors for Heart Failure as described in the table below
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Measuring Cardiac Output for wireless transmission as per discharge guideline | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vijay, MD, MS, FACC, Principal Investigator — Scottsdale Healthcare
Locations (1):
- Scottsdale Cardiovascular Center, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. BMJ. 2007 May 5;334(7600):942. doi: 10.1136/bmj.39156.536968.55. Epub 2007 Apr 10. PMID 17426062
- [Background] Inglis SC, Clark RA, McAlister FA, Ball J, Lewinter C, Cullington D, Stewart S, Cleland JG. Structured telephone support or telemonitoring programmes for patients with chronic heart failure. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007228. doi: 10.1002/14651858.CD007228.pub2. PMID 20687083
- [Result] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- See also: Evaluate Heart Failure Patients With Specially Designed Patient Adherence and Monitoring Software on Standard Mobile Devices (REMOTE-HF-1) — http://clinicaltrials.gov/show/NCT01430936